CLINICAL TRIAL: NCT05173506
Title: CHICA-CN Evaluation - Evaluation of a Computer Decision Support System in Child Neurology
Brief Title: Child Health Improvement Through Computer Automation - Child Neurology (CHICA-CN) Evaluation
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Norton Healthcare (Other); Indiana University (Other); Child Neurology Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00078610
Record Dates: First submitted 2021-11-17; First posted 2021-12-30 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-08

CONDITIONS: Neurologic Disorder
Keywords: Quality of Care; Child Health Improvement
MeSH Terms: conditions — Nervous System Diseases | interventions — Physicians

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adolescent Depression Screening: * > 3 visits to clinic
  * Diagnosis of epilepsy - International Classification of Diseases, Tenth Revision - Epilepsy and recurrent seizures (ICD-10:G40)
  * Age > 12 years at last visit (before CHICA-CN)
  Computer assistant depression screening and management
  Interventions: Other: Computer decision support for physician
- Genetic Testing: * > 3 visits to clinic
  * Diagnosis of global developmental delay - International Classification of Diseases, Tenth Revision - autistic disorder (ICD-10: F84)
  * Age < 6 years at last visit (before CHICA-CN)
  Computer reminders to test for genetic disorders
  Interventions: Other: Computer decision support for physician
- Rescue seizure therapy: * > 3 visits to clinic
  * Diagnosis of epilepsy - International Classification of Diseases, Tenth Revision - Epilepsy and recurrent seizures (ICD-10: G40)
  * Age < 18 years at last visit (before CHICA-CN)
  Computer reminders to prescribe and adjust rescue anti-seizure medications
  Interventions: Other: Computer decision support for physician
- Adolescent Transition: * > 3 visits to clinic
  * Age > 13 years at last visit (before CHICA-CN)
  Computer supported screening and counseling regarding transition to adult care
  Interventions: Other: Computer decision support for physician

INTERVENTIONS:
Other: Computer decision support for physician — The Child Health Improvement through Computer Automation - Child Neurology (CHICA-CN) system will screen patients for needed services and provide reminders to physicians to provide the needed services.

SUMMARY:
The study will evaluate a computer decision support system for child neurology, Child Health Improvement through Computer Automation - Child Neurology (CHICA-CN) using patient chart review, family phone surveys, and physician interviews in a before-after study design.

DETAILED DESCRIPTION:
(CHICA-CN) Child Health Improvement through Computer Automation - Child Neurology is software that works with the electronic health record (EHR) to improve the efficiency and quality of care in the outpatient setting. Built in partnership with the Child Neurology Foundation, CHICA's guidance is based on authoritative guidelines from the American Academy of Neurology and others. The plan is to implement CHICA-CN in the Child Neurology Clinics at Wake Forest Baptist Health. To evaluate CHICA-CN the proposal is to look at data derived from three sources:

1. Chart Review to evaluate quality of care based on measures derived from four algorithms developed from American Academy of Neurology quality measures and typically documented in the medical record. This will be a before-after study design in which measurements will be obtained before and after the installation of CHICA-CN.
2. Parent Phone Surveys to Document the parent experience in terms of physician-patient communication, parent engagement, and satisfaction with use of the patient facing tablet interface. These data will be collected from families of patients identified for the chart review after the intervention.
3. Physician user satisfaction measures, including perceived value of the system and ease of use in general and as regards individual clinical issues. Surveys will be administered to physicians and clinic staff who used CHICA-CN.

ELIGIBILITY:
Inclusion Criteria:

* Must be patients in the participating clinical practices meeting inclusion criteria for one of the four cohorts

Exclusion Criteria:

* N/A

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children under 18 years of age who attend one of two participating child neurology clinics who qualify for one of the four cohorts and who have at least three visits to that clinic and at least one visit during the study period
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Chart Abstraction Outcomes - Transitions of Care | Visits will be extracted for the year before implementation of CHICA-CN and for a one year period after implementation of CHICA-CN
  Transitions of Care - the number of charts that document that the service was provided divided by the number of charts reviewed
Chart Abstraction Outcomes - Rescue Seizure Therapy for Children with Epilepsy | Visits will be extracted for the year before implementation of CHICA-CN and for a one year period after implementation of CHICA-CN
  Rescue Seizure Therapy for Children with Epilepsy - the number of charts that document that the service was provided divided by the number of charts reviewed
Chart Abstraction Outcomes - Genetic Testing for Global Developmental Delay | Visits will be extracted for the year before implementation of CHICA-CN and for a one year period after implementation of CHICA-CN
  Genetic Testing for Global Developmental Delay - the number of charts that document that the service was provided divided by the number of charts reviewed
Chart Abstraction Outcomes - Adolescent Depression Screening | Visits will be extracted for the year before implementation of CHICA-CN and for a one year period after implementation of CHICA-CN
  Adolescent Depression Screening - the number of charts that document that the service was provided divided by the number of charts reviewed
Physician-patient communication Survey Score | Eligible patients will be identified as they have encounters, starting 6 months after implementation of CHICA-CN and continuing for 12 months, assessed for the identified visit, within 2 weeks of the visit
  Communication subscale of the Ambulatory Care Experiences (ACE) Survey - includes 4 items like "How often did your personal doctor explain things in a way that was easy to understand" or "How would you rate your personal doctor's knowledge of your medical history." - Single score (0-12), higher score indicates better communication.
Patient engagement Survey Score | Eligible patients will be identified as they have encounters, starting 6 months after implementation of CHICA-CN and continuing for 12 months, assessed for the identified visit, within 2 weeks of the visit
  Patient Activation Measure Short Form (PAM) - 13 item scale assesses whether the parent believes an active role in the child's care is important; if the parent has the confidence and knowledge to take action, e.g., medications, bringing concerns to the provider; if the parent has taken action, e.g., lifestyle changes, to improve child's health; and whether the parent stays on course under stress, e.g., being able to handle child's health condition at home. 13 items, single score (0-39), higher score indicates greater patient/parent engagement.
Physician Satisfaction Survey | After one year of of clinicians using CHICA-CN
  Clinician user satisfaction measures, including perceived value of the system and ease of use in general and as regards individual clinical issues. Surveys will be administered to physicians and clinic staff who used CHICA-CN. The survey includes a series of statements with which the respondent will mark their level of agreement on a Likert scale. There is no summary score, but we will calculate and report a mean, median, and range for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn M Martindale, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.